CLINICAL TRIAL: NCT06389968
Title: Lichtstimulation Zur Verbesserung Der Sehleistung Bei Patientinnen Und Patienten Mit Multipler Sklerose Nach Sehnerventzündung
Brief Title: Light Stimulation to Improve Visual Function After Optic Neuritis in Persons with Multiple Sclerosis
Acronym: ONSTIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2023-491-S-KH
Record Dates: First submitted 2024-04-22; First posted 2024-04-29 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Optic Neuritis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Optic Neuritis

STUDY DESIGN:
Intervention Model Description: sham-controlled
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Light stimulation (Experimental): Experimental light stimulation (3 colors at 20 Hertz each for 80 seconds twice a day).
  Interventions: Device: Light stimulation
- Sham light stimulation (Sham Comparator): Sham light stimulation (white screen for 80 seconds twice a day).
  Interventions: Device: Sham light stimulation

INTERVENTIONS:
Device: Light stimulation — see arm description
  Arms: Light stimulation
Device: Sham light stimulation — see arm description
  Arms: Sham light stimulation

SUMMARY:
The aim of this monocentric randomized controlled intervention study is to improve visual function in persons with multiple sclerosis following optic neuritis (neuritis nervi optici) by means of a light stimulation.

In the treatment arm, two 80-second light stimulations are to be administered daily for 12 days in 25 persons with multiple sclerosis following recent optic neuritis (1-3 months). For the standardized application of light stimulation in the sense of standardized training, the light stimulation is to be carried out by watching a generated flicker video on a mobile phone. In a sham-intervened control group (sample size 25), the spontaneous course after optic neuritis will be recorded in parallel. Intensive neuronal stimulation of the visual pathway will be used to stimulate regenerative processes, which will be recorded by means of changes in high-contrast visual acuity (primary endpoint). Secondary endpoints are changes in a colored-contrast test, in 2.5% low contrast visual acuity, the peak conduction latency of visual evoked potentials, and retinal layer thicknesses and vessel densities measured in optical coherence tomography and optical coherence tomorgraphic angiography. These physiological parameters should help to understand the underlying processes of a potentially altered visual performance.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing remitting multiple sclerosis or clinically isolated syndrome or no indication of chronic inflammatory central nervous system disease
* Age 18-60 years
* Optic neuritis within 1-3 months

Exclusion Criteria:

* Epilepsy
* Light-triggered migraine
* Insufficient vision correction
* Retinal disease (glaucoma, macular edema, macula degeneration, ...)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
High contrast visual sensitivity | before intervention, directly after the first stimulation, after 12 days of training (stimulation) as 24 hour retention, and at 22 days post-intervention (retention)
  Visual resolution with Sloan chart

SECONDARY OUTCOMES:
Low contrast visual sensitivity | before intervention, directly after the first stimulation, after 12 days of training (stimulation) as 24 hour retention, and at 22 days post-intervention (retention)
  Sloan chart at 2.5%
Visually evoked potentials | before intervention, directly after the first stimulation, after 12 days of training (stimulation) as 24 hour retention, and at 22 days post-intervention (retention)
  Visually evoked potential
Optical coherence tomography | before intervention, directly after the first stimulation, after 12 days of training (stimulation) as 24 hour retention, and at 22 days post-intervention (retention)
  Optical coherence tomography
Optical coherence tomographic angiography | before intervention, directly after the first stimulation, after 12 days of training (stimulation) as 24 hour retention, and at 22 days post-intervention (retention)
  Optical coherence tomographic angiography
Color contrast | before intervention, directly after the first stimulation, after 12 days of training (stimulation) as 24 hour retention, and at 22 days post-intervention (retention)
  Color contrast threshold (3 colors)

CONTACTS AND LOCATIONS:
Locations (1):
- Technical University of Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No